CLINICAL TRIAL: NCT02958306
Title: Evaluation of the Effect of Platelet Rich Plasma (PRP) on the Esthetic Outcome and Scar Formation of Unilateral Cleft Lip Repair by Modified Millard Cheiloplasty: A Randomized Clinical Trial
Brief Title: Effect of Platelet Rich Plasma (PRP) on the Esthetic Outcome and Scar Formation of Unilateral Cleft Lip Repair
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SMohasin
Record Dates: First submitted 2016-11-03; First posted 2016-11-08 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Unilateral Cleft Lip
Keywords: cleft lip repair; cheiloplasty; PRP; platelet rich plasma

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- platelet rich plasma (Experimental): autologous blood product
  Interventions: Biological: platelet rich plasma
- no platelet rich plasma (No Intervention): control

INTERVENTIONS:
Biological: platelet rich plasma — PRP is a portion of the plasma fraction of autologous blood, having a platelet concentration above baseline values
  Other Names: PRP
  Arms: platelet rich plasma

SUMMARY:
The purpose of this study is to evaluate effect of platelet rich plasma on scar formation of unilateral cleft lip repair.

DETAILED DESCRIPTION:
PRP is a portion of the plasma fraction of autologous blood, having a platelet concentration above baseline values. PRP is made by centrifugation of whole blood (drawn from a peripheral vein and stored in an acid citrate dextrose solution A (ACD-A) anticoagulant), which separates the various components of blood by their specific weight and increases the concentration of platelets.

Platelets are a rich source of the complex group of proteins called growth factors (GFs) involved in natural wound healing and in regeneration of injured tissues. GFs are active signals for attracting stem cells into the site of injury and triggering proliferation of these cells. PRP limit inflammation, interacting with macrophages to improve tissue healing and regeneration, promote new capillary growth, and accelerate epithelialization. Platelets in PRP also play a role in host defense mechanism at the wound site by producing signaling proteins that attract macrophages; PRP also may contain a small number of leukocytes that synthesize interleukins as part of a non-specific immune response. Previous studies of PRP have demonstrated antimicrobial activity against Escherichia coli, Staphylococcus aureus, including methicillin-resistant Staphylococcus aureus, Candida albicans, and Cryptococcus neoforma. So, PRP is effective in soft tissue healing, having no side effect and showed excellent healing score in skin wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nonsyndromic cleft lip
* Primary, unilateral, complete or incomplete cleft lip
* Patient's age younger than six months
* Lip repair performed by one craniofacial surgeon
* Completeness of medical records including preoperative and postoperative photographs at approximately 6 months after surgery

Exclusion Criteria:

* Patients with syndromic cleft lip
* Secondary lip treatment (previous operated cases)
* Bilateral cleft lip
* Patient older than six months
* Associated Cardiac anomalies
* Any systemic condition

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
scar width | 6 months
  scar width through orbicularis oris muscle by ultrasonography
scar width | 6months
  scar width at skin surface via photograph

SECONDARY OUTCOMES:
vancouver scar scale | 6 months
  VSS has four parameters, including vascularity, pigmentation, thickness, and pliability giving a range of 0 to 13 in the total score with 0 representing normal skin

OTHER OUTCOMES:
Philtral ridge length symmetry index | 6months
  Philtral ridge length was measured on the non-cleft side and a correspondent length on the reconstructed cleft side from nasal sill to the peak of Cupid's bow . Philtral ridge symmetry index was calculated as follow:- (Cleft side component value)/(Non clefted side component value)×100

CONTACTS AND LOCATIONS:
Overall Officials: basma G mousa, professor, Study Director — Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided